CLINICAL TRIAL: NCT00816231
Title: Drug /Cue Interactions In Alcohol-Tobacco Comorbidity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MCC-14671
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Nicotine Dependence
Keywords: Prevention Intervention; Alcohol; Tobacco; Nicotine; Craving; Cue Reactivity; Cross Cue Reactions
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Products; Alcoholic Beverages

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Alcohol and Nicotine Group (Experimental): Alcohol and Nicotine Drug/Cue Interactions
  Interventions: Behavioral: Tobacco; Other: Alcoholic Beverage
- Alcohol Only Group (Active Comparator): Alcohol Only Drug/Cue Interactions
  Interventions: Other: Alcoholic Beverage; Other: Placebo
- Nicotine Only Group (Active Comparator): Nicotine Only Drug/Cue Interactions
  Interventions: Behavioral: Tobacco; Other: Placebo
- Placebo and Placebo Group (Placebo Comparator): Placebo Only Drug/Cue Interactions
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Tobacco — Five research sessions. Session 1: Questionnaires, interviews, computer task, medical evaluation. Sessions 2 - 5: Lab Sessions involving tobacco with brief summary at the end of the last session.
  Arms: Alcohol and Nicotine Group; Nicotine Only Group
Other: Alcoholic Beverage — Five research sessions. Session 1: Questionnaires, interviews, computer task, medical evaluation. Sessions 2 - 5: Lab Sessions involving and alcohol with brief summary at the end of the last session.
  Arms: Alcohol Only Group; Alcohol and Nicotine Group
Other: Placebo — Five research sessions. Session 1: Questionnaires, interviews, computer task, medical evaluation. Sessions 2 - 5: Lab Sessions involving placebo with brief summary at the end of the last session.
  Arms: Alcohol Only Group; Nicotine Only Group; Placebo and Placebo Group

SUMMARY:
The purpose of this study is to determine how people react to different combinations of alcohol and nicotine.

DETAILED DESCRIPTION:
The present project will improve and expand upon previously published work in several ways. First, Study 1 will assess reactivity to alcohol and smoking cues in the same session. Second, both studies will include within-subjects design factors to manipulate alcohol and nicotine intake, as well as cue types. Third, craving indices will represent three important response domains: subjective, physiological, and behavioral (e.g., Niaura et al., 1991). Fourth, each study will evaluate a range of drinkers and smokers, which will provide maximal information concerning influences on alcohol and smoking cue reactivity across various subject populations. The proposed studies are not only important from a theory development perspective, but they will provide an excellent foundation for future laboratory-based and clinical research.

ELIGIBILITY:
Inclusion Criteria:

* English speaking persons who exhibit a range of alcohol consumption and smoking patterns.
* Signed written consent form.

Exclusion Criteria:

* Females who are pregnant, nursing, or not using effective methods of birth control will be excluded from participating.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2006-05-08 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Psychophysiological Reactivity Assessment | approximately 5 weeks per participant
  To assess cravings and psychophysiological reactivity elicited by alcohol, smoking, and neutral cues following acute intake of alcohol and nicotine among individuals across a broad range of alcohol and cigarette use patterns (Study 1).

SECONDARY OUTCOMES:
Alcohol Self-administration Assessment | approximately 5 weeks per participant.
  To assess alcohol self-administration upon exposure to alcohol or smoking-related cues following acute intake of alcohol, nicotine, or both drugs among individuals across a broad range of alcohol and cigarette use patterns (Study 2).

CONTACTS AND LOCATIONS:
Overall Officials: David Drobes, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States